CLINICAL TRIAL: NCT06462521
Title: Cold Snare Piecemeal Resection vs Cold Snare Endoscopic Mucosal Resection: A RandomizeD Trial IN Colorectal Adenomas 10-19mm and Serrated Lesions ≥ 10mm (CARDINAL Study)
Brief Title: Cold Snare Piecemeal Resection vs Cold Snare Endoscopic Mucosal Resection
Acronym: CARDINAL
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Rush University Medical Center (Other); University of Colorado, Denver (Other); John D. Dingell VA Medical Center (U.S. Federal Agency); White River Junction Veterans Affairs Medical Center (U.S. Federal Agency); University of Kansas Medical Center (Other); Vancouver Coastal Health (Other Government); Université de Montréal (Other); University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, John J. Guardiola, Assistant Professor of Clinical Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20831
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-09

CONDITIONS: Colon Cancer; Colon Polyp; Colon Adenoma; Serrated Polyp
Keywords: Polyp Resection; Cold Snare; Cold Endoscopic Mucosal Resection (Cold EMR); Cold Snare Piecemeal Resection (CSPR); Colonoscopy
MeSH Terms: conditions — Colonic Neoplasms; Colonic Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold Snare Piecemeal Resection (CSPR) (Experimental): Conventional adenomas sized 10-19mm or serrated lesions 10mm or larger found during colonoscopy will be removed using CSPR technique.
  Interventions: Procedure: Cold Snare Piecemeal Resection (CSPR)
- Cold Snare Endoscopic Mucosal Resection (Cold EMR) (Experimental): Conventional adenomas sized 10-19mm or serrated lesions 10mm or larger found during colonoscopy will be removed using Cold EMR technique.
  Interventions: Procedure: Cold Snare Endoscopic Mucosal Resection (Cold EMR)

INTERVENTIONS:
Procedure: Cold Snare Piecemeal Resection (CSPR) — Qualifying polyps randomized to Cold Snare Piecemeal Resection (CSPR) will be removed using cold snare techniques (no electrocautery, no submucosal injection.)
  Arms: Cold Snare Piecemeal Resection (CSPR)
Procedure: Cold Snare Endoscopic Mucosal Resection (Cold EMR) — Qualifying polyps randomized to Cold Snare Endoscopic Mucosal Resection (Cold EMR) will be removed using cold snare techniques (no electrocautery, with submucosal injection.)
  Arms: Cold Snare Endoscopic Mucosal Resection (Cold EMR)

SUMMARY:
The study will compare the use of cold snare piecemeal resection (CSPR) vs cold endoscopic mucosal resection (Cold EMR). The study will include two cohorts: one cohort for conventional adenomas 10-19mm in size and one cohort for serrated lesions 10mm or larger.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Presenting for a screening, surveillance, diagnostic, or therapeutic colonoscopy
3. Found to have:

   * a sessile serrated lesion or hyperplastic polyp ≥ 10 mm during procedure (Serrated Cohort) or
   * a 10-19 mm conventional adenoma during procedure (Adenoma Cohort)
4. Ability to provide informed consent

Exclusion Criteria:

1. Pedunculated or semi-pedunculated polyps (as defined by Paris Classification type Ip or Isp)
2. Polyps confirmed to be anything other than:

   * sessile serrated lesion or hyperplastic polyp on histologic diagnosis (Serrated Cohort) or
   * conventional adenoma on histologic diagnosis (Adenoma Cohort)
3. Patients with Ulcerative Colitis or Crohn's disease
4. Polyps with features suggestive of submucosal invasion
5. Polyps that are not able to be removed endoscopically due to location (e.g. extending into appendiceal orifice or diverticulum)
6. Patients with a known or suspected diagnosis of any of the following polyposis syndromes with known genetic mutations:

   * Familial Adenomatous Polyposis Syndrome
   * MUTYH associated Polyposis Syndrome
   * Juvenile Polyposis Syndrome
   * Cowden's Syndrome
   * Peutz-Jeghers Syndrome
7. Subjects whose colonoscopy procedure is not able to be completed due to bowel prep precluding polyp identification.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 570 (Estimated)
Dates: Start 2024-09-06 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Resection (Central Post-Resection Biopsies) | 1 day
  Efficacy of resection will be assessed by biopsies in four or six quadrants of the perimeter of the defect post-resection and two biopsies from the center of the defect post-resection. Comparison of the biopsy pathology results for polyps removed by Cold EMR vs CSPR.
Efficacy of Resection (Peripheral Post-Resection Biopsies) | 1 day
  Efficacy of resection will be assessed by biopsies in four or six quadrants of the perimeter of the defect post-resection and two biopsies from the center of the defect post-resection. Comparison of the biopsy pathology results for polyps removed by Cold EMR vs CSPR.

SECONDARY OUTCOMES:
Polyp Resection Time | 1 day
  The time it takes to remove the polyp completely
Resection Preparation Time | 1 day
  The time it takes to prepare for polyp removal
Total Procedure Time | 1 day
  The total time it takes to complete the colonoscopy procedure
Adverse Events | 30 Days
  The number of complications for each randomization arm during and after the procedure
Rate of Recurrence at First Surveillance Colonoscopy for Polyps ≥ 20mm | At first surveillance colonoscopy, typically 6 months to 12 months
  The recurrence rate of serrated lesions ≥ 20mm measured at the first follow-up colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: John J Guardiola, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data may be shared in the future upon request per PI discretion.

REFERENCES:
- [Background] Kaltenbach T, Anderson JC, Burke CA, Dominitz JA, Gupta S, Lieberman D, Robertson DJ, Shaukat A, Syngal S, Rex DK. Endoscopic Removal of Colorectal Lesions-Recommendations by the US Multi-Society Task Force on Colorectal Cancer. Gastroenterology. 2020 Mar;158(4):1095-1129. doi: 10.1053/j.gastro.2019.12.018. Epub 2020 Feb 11. No abstract available. PMID 32122632
- [Background] von Renteln D, Djinbachian R, Benard F, Barkun AN, Bouin M, Bouchard S, Deslandres E, Panzini B, Sidani S, Leduc R, Jobse BC, Pohl H. Incomplete resection of colorectal polyps of 4-20 mm in size when using a cold snare, and its associated factors. Endoscopy. 2023 Oct;55(10):929-937. doi: 10.1055/a-1978-3277. Epub 2022 Nov 14. PMID 36377124
- [Result] McWhinney CD, Vemulapalli KC, El Rahyel A, Abdullah N, Rex DK. Adverse events and residual lesion rate after cold endoscopic mucosal resection of serrated lesions >/=10 mm. Gastrointest Endosc. 2021 Mar;93(3):654-659. doi: 10.1016/j.gie.2020.08.032. Epub 2020 Sep 3. PMID 32891621
- [Result] Rex DK, Anderson JC, Pohl H, Lahr RE, Judd S, Antaki F, Lilley K, Castelluccio PF, Vemulapalli KC. Cold versus hot snare resection with or without submucosal injection of 6- to 15-mm colorectal polyps: a randomized controlled trial. Gastrointest Endosc. 2022 Aug;96(2):330-338. doi: 10.1016/j.gie.2022.03.006. Epub 2022 Mar 12. PMID 35288147
- [Result] Kimoto Y, Sakai E, Inamoto R, Kurebayashi M, Takayanagi S, Hirata T, Suzuki Y, Ishii R, Konishi T, Kanda K, Negishi R, Takita M, Ono K, Minato Y, Muramoto T, Ohata K. Safety and Efficacy of Cold Snare Polypectomy Without Submucosal Injection for Large Sessile Serrated Lesions: A Prospective Study. Clin Gastroenterol Hepatol. 2022 Feb;20(2):e132-e138. doi: 10.1016/j.cgh.2020.10.053. Epub 2020 Nov 2. PMID 33152541
- [Result] Mangira D, Raftopoulos S, Vogrin S, Hartley I, Mack A, Gazelakis K, Nalankilli K, Trinh A, Metz AJ, Appleyard M, Grimpen F, Elliott T, Brown G, Moss A. Effectiveness and safety of cold snare polypectomy and cold endoscopic mucosal resection for nonpedunculated colorectal polyps of 10-19 mm: a multicenter observational cohort study. Endoscopy. 2023 Jul;55(7):627-635. doi: 10.1055/a-2029-9539. Epub 2023 Feb 7. PMID 36750222
- [Result] Gupta S, Lieberman D, Anderson JC, Burke CA, Dominitz JA, Kaltenbach T, Robertson DJ, Shaukat A, Syngal S, Rex DK. Recommendations for Follow-Up After Colonoscopy and Polypectomy: A Consensus Update by the US Multi-Society Task Force on Colorectal Cancer. Gastroenterology. 2020 Mar;158(4):1131-1153.e5. doi: 10.1053/j.gastro.2019.10.026. Epub 2020 Feb 7. No abstract available. PMID 32044092